CLINICAL TRIAL: NCT03980600
Title: Suitability of Nanocellulose Wound Dressing for the Treatment of Skin Graft Donor Sites
Brief Title: NFC Dressing for Skin Graft Donor Sites
Acronym: FibDexHBC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: UPM-Kymmene Corporation (Industry)
Collaborators: University of Helsinki (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HUS/1166/2016
Record Dates: First submitted 2019-05-23; First posted 2019-06-10 (Actual); Last update posted 2019-06-10 (Actual); Status verified 2019-06

CONDITIONS: Skin Transplantation

STUDY DESIGN:
Intervention Model Description: Single center clinical investigation with patients selected by the clinicians. The donor sites were treated and compared intra-individually in the same patients.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Donor site treatment with NFC dressing/FibDex® (Experimental): Patients requiring skin graft donor site treatment were enrolled in the investigation. Patients were selected based on clinical evaluation by a plastic surgeon.
  Of the total 33 patients enrolled in the study, nine patients were treated during the optimization phase with experimental NFC dressing Types 1-3. The remaining 24 patients were treated with the final product Type 4 (FibDex®). The mean age of patients treated with NFC dressing/FibDex® was 50 ± 18 years, in the range of 21-74 years.
  Suprathel® was used to treat donor sites in the same patients as a reference material. During the optimization phase, Suprathel was intra-individually compared with NFC dressing types 1-3 in five patients out of nine. From the remaining 24 patients, Suprathel was intra-individually compared with FibDex® in 17 patients.
  Interventions: Device: FibDex wound dressing; Device: NFC wound dressing Types 1-3; Device: Suprathel (comparator)

INTERVENTIONS:
Device: FibDex wound dressing — Treatment of donor sites of 24 patients with the dressing Type 4 (final product i.e. FibDex) until the self-detachment of the wound dressing i.e. epithelialization
  Other Names: NFC wound dressing
Device: NFC wound dressing Types 1-3 — Treatment of donor sites of 9 patients with the NFC dressing's (proto)Types 1-3 until the self-detachment of the wound dressing i.e. epithelialization
Device: Suprathel (comparator) — Treatment of donor sites of 22 patients with Suprathel dressing, which was used as a reference (comparator) product, until the self-detachment of the wound dressing i.e. epithelialization

SUMMARY:
The aim of this single center clinical investigation was to optimize nanofibrillar cellulose (NFC) wound dressing and to investigate final product FibDex in the treatment of split thickness skin graft donor sites. Performance of NFC dressings Type 1, Type 2, Type 3 and Type 4 (final product, FibDex) was compared with that of Suprathel®.

DETAILED DESCRIPTION:
The aim of this study was to investigate the suitability of FibDex for the treatment of skin graft donor sites. The study results will help to 1) ensure that the performance of the study product corresponds to product definition, 2) estimate the study product suitability for use and 3) determine the potentially emerging adverse effects of the study product.

During the clinical investigation the study product has been in normal use, as defined by the manufacturer in the intended use. Those members of the study team who work at the study location gave their assessment on the suitability of the NFC dressing for treating the patients using their clinical assessment and experience.

The NFC dressing was used during the study to protect the skin graft donor sites, and its effect on the skin graft donor site healing was compared to Suprathel® (PolyMedics Innovations GmbH, Germany). Suprathel® is the most commonly used skin graft donor site material for the treatment of large burns at the Helsinki Burn Centre. Suprathel® has similar indications and applications as the NFC dressing.

The clinical study was performed according to the Clinical Investigation of medical devices for human subjects, good clinical practice (ISO 14155:2011) at Helsinki Burn Centre, Helsinki University Hospital, Finland. The study was approved by the Research Ethics Committee at the Helsinki University Hospital (99/13/03/02/2014 and HUS/1166/2016), and enrolled burn patients or patients requiring skin graft donor site treatment with exclusion criteria of pregnancy and age under 18 or over 75 years. Subjects or their legal representatives were informed of procedures and provided written informed consent. Altogether 24 patients were treated with FibDex, having a comparison to Suprathel® with 17 patients. It was hypothesized that, due to the inherent characteristics of NFC, treatment of donor sites with FibDex would expedite wound healing.

A Zimmer® air dermatome (Zimmer Inc., USA) was used to harvest 6/1000 inch (0.15 mm)-12/1000 inch (0.30 mm) thick split-thickness skin grafts. The separate donor sites were covered with FibDex or with FibDex and Suprathel® except in one patient whose single donor site was divided into two parts and treated with both dressings. Experimental dressings that were left in place for the entire treatment period were covered by Jelonet® (Smith & Nephew, UK) and fixed with staples. When compared to Suprathel®, anatomically equivalent areas were chosen for donor sites. The dressings were randomly selected for treatment of each donor site.

The healing time of the donor site was determined as the self-detachment day of FibDex or Suprathel® + Jelonet® dressings. Both donor site materials behave similarly detaching from the wound bed when new epithelium is regenerated. Postoperatively, the experimental dressings on skin graft donor sites were checked by visual observation when changing the overlaying dressings at interval of a few days on average on postoperative days (POD) 4, 7, 10, 14, 20 and 28, or when clinically relevant (±1-3 days), until self-detachment. During observations, skin quality, the epithelialization percentage of the donor site skin and the possible adverse effects were evaluated by a plastic surgeon. In addition, subjective pain experience was questioned from the patients using scale 0-10 (0 representing no pain and 10 the worst possible pain). Donor sites and wound dressings were photographed during the examinations throughout the clinical study period. Skin elasticity, viscoelasticity and TEWL were measured after discharge, one and six months postoperatively. In addition, scar quality was evaluated using the POSAS that was translated to Finnish but not validated in Finnish language. The POSAS consists of two numerical scales, the patient and the observer scar assessment scale that scores six parameters on a 10-point rating scale, in which the highest score represents the worst imaginable scar.

Elasticity, viscoelasticity and TEWL were measured from patients' epithelialized skin treated with FibDex dressing or Suprathel® during follow up examination at one and six months after commencement of the treatments using DermaLab® Skinlab COMBO (Cortex Technology, Denmark), which is a reliable instrument for objective measurements of skin elasticity and TEWL. The elasticity of the skin was assessed in terms of elastic modulus and viscoelasticity. TEWL was expressed as g/m2/h to assess the epidermal barrier function. Transepidermal water loss increases when the skin barrier is damaged and is therefore an important parameter to evaluate the efficiency of the human skin barrier. For measurements, a single (in case of TEWL measurement) or 4-5 (in case of elasticity measurements) successive readings were taken at the same site. Control measurements were taken on healthy, not operated skin of the same subject at equal location.

ELIGIBILITY:
Inclusion Criteria:

- Patients with a need of skin graft donor site treatment under 10 % of the total body area

Exclusion Criteria:

* Pregnancy
* Age under 18
* Age over 75

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2015-02-16 (Actual); Primary Completion 2018-01-08 (Actual); Study Completion 2018-09-19 (Actual)

PRIMARY OUTCOMES:
Wound healing time | Postoperative day (POD) as a checkpoint :14 days
  The healing time of the donor site was determined as the self-detachment day of the dressing that was checked by visual observation at interval of a few days until self-detachment.
Wound healing time | Postoperative day (POD) as a checkpoint: 1 month
  The healing time of the donor site was determined as the self-detachment day

SECONDARY OUTCOMES:
Subjective pain | On postoperative day (POD) 10-15, 1 month and 6 months review
  Subjective pain experience was questioned from the patients using scale 0-10 (0 representing no pain and 10 the worst possible pain).
Epithelialization | Postoperative day (POD) 14, 1 month, 6 months
  Percentage of epithelialization was evaluated by visual observation by a plastic surgeon.
Scar quality | 1 month and 6 months postoperatively
  Appearance of scar was evaluated using the Patient and Observer Scar Assessment Scale (POSAS) consisting of two numerical scales, the patient and the observer scar assessment scale that scores six parameters (vascularity, pigmentation, thickness, relief, pliability and surface area on the observer scale, and pain, itching, color, pliability, thickness and relief on the patient scale) on a 10-point rating scale (0-10), in which the highest score represents the worst imaginable scar.
Skin elasticity | 1 month and 6 months postoperatively
  Elasticity was measured from patients' epithelialized donor site after commencement of the treatments using DermaLab® Skinlab COMBO instrument. The elasticity of the skin was assessed in terms of elastic modulus. For measurements, 4-5 successive readings were taken at the same site. Control measurements were taken on healthy, not operated skin of the same subject at equal location.
Transepidermal water loss (TEWL) | 1 month and 6 months postoperatively
  TEWL was measured from patients' epithelialized donor site after commencement of the treatments using DermaLab® Skinlab COMBO instrument. TEWL was expressed as g/m2/h to assess the epidermal barrier function. Transepidermal water loss values increase when the skin barrier is damaged. For measurements, a single successive reading was taken. Control measurements were taken on healthy, not operated skin of the same subject at equal location.
Viscoelasticity | 1 month and 6 months postoperatively
  Viscoelasticity was measured from patients' epithelialized donor site after commencement of the treatments using DermaLab® Skinlab COMBO instrument, and expressed as megapascals (MPa). For measurements, 4-5 successive readings were taken at the same site. Control measurements were taken on healthy, not operated skin of the same subject at equal location.

CONTACTS AND LOCATIONS:
Overall Officials: Jyrki Vuola, MD, PhD, Principal Investigator — Helsinki Burn Centre, Helsinki University Hospital
Locations (1):
- Helsinki Burn Centre, Department of Plastic Surgery, Helsinki University Hospital, Espoo, Finland

IPD SHARING:
Plan to Share IPD: No